CLINICAL TRIAL: NCT03645590
Title: Stroke Ready - Optimizing Acute Stroke Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Lesli Skolarus, Associate Professor of Neurology, University of Michigan
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: U01MD010579 (NIH); U01MD010579 (NIH)
Record Dates: First submitted 2017-03-23; First posted 2018-08-24 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Stroke, Acute; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Stroke Ready is a stepped wedge design to be delivered to each of the four Flint community quadrants over the course of 2 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stroke Ready Community intervention (Experimental): We divided the Flint community into four quadrants. We will focus our workshops and posters on one quadrant, but not exclusively, moving quadrants every 6 months over the course of two years.
  Interventions: Behavioral: Stroke Ready

INTERVENTIONS:
Behavioral: Stroke Ready — Stroke Ready community intervention consists of peer facilitated educational workshops, stroke music video, and mass media campaign including print materials (e.g. posters, brochure), health promotion mailers, radio/Television public health service announcements, and the Stroke Ready website and Facebook page.

SUMMARY:
The study aims to increase acute stroke treatment rates in Flint, Michigan through a two-pronged approach of hospital and community level interventions. It also aims to inform future stroke preparedness interventions by exploring the relative importance of hospital optimization and community interventions.

ELIGIBILITY:
Inclusion criteria:Adult stroke patients who presented to one of three hospitals in the Flint community.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5970 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Acute stroke treatment rate (tPA) | Time frame: 11 years of data will be reviewed
  Acute stroke treatment rate - community wide. Retrospective data captured through medical record review

SECONDARY OUTCOMES:
Number of emergency department arrivals by ambulance | Time frame: 11 years of data will be reviewed
  Optimize community for acute stroke (community level)--retrospective data captured through medical record review

CONTACTS AND LOCATIONS:
Overall Officials: Lesli Skolarus, MD, Principal Investigator — University of Michigan
Locations (1):
- Flint Communiy, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Robles MC, Springer MV, Corches CL, Burke JF, Lin CC, Oliver A, Skolarus LE. Stroke Ready Very Brief Intervention Improves Immediate Postintervention Stroke Preparedness. Circ Cardiovasc Qual Outcomes. 2020 Dec;13(12):e006643. doi: 10.1161/CIRCOUTCOMES.120.006643. Epub 2020 Nov 26. No abstract available. PMID 33238728
- [Derived] Skolarus LE, Sales AE, Zimmerman MA, Corches CL, Landis-Lewis Z, Robles MC, McBride AC, Rehman N, Oliver A, Islam N, Springer MV, O'Brien A, Bailey S, Morgenstern LB, Meurer WJ, Burke JF. Stroke Ready: a multi-level program that combines implementation science and community-based participatory research approaches to increase acute stroke treatment: protocol for a stepped wedge trial. Implement Sci. 2019 Mar 7;14(1):24. doi: 10.1186/s13012-019-0869-3. PMID 30845958